CLINICAL TRIAL: NCT00347828
Title: Prospective Study Comparing the Effectiveness of Zymar and Vigamox for Preoperative Antibiotic Sterilization of the Ocular Surface After Loading Dose
Brief Title: Effectiveness Study of Zymar Versus Vigamox for Preoperative Sterilization of the Ocular Surface After Loading Dose
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ophthalmic Consultants of Boston (Other)
Collaborators: Allergan (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: Allergan/Z101
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2006-07-04 (Estimated); Status verified 2006-06

CONDITIONS: Eye Infection; Infection
Keywords: Antibiotic prophylaxis; Vigamox; Moxifloxacin; Zymar; Gatifloxacin; Preoperative antibiotic; Eye infection
MeSH Terms: conditions — Eye Infections; Infections

INTERVENTIONS:
Drug: Moxifloxacin ophthalmic solution 0.5%
Drug: Gatifloxacin ophthalmic solution 0.3%

SUMMARY:
The purpose of this study is to analyze the effect of Zymar and Vigamox on ocular surface bacteria. We believe that Zymar will eradicate more ocular surface bacteria than Vigamox.

DETAILED DESCRIPTION:
Topical antibiotics are frequently used before surgical procedures with the intent of targetting and reducing the number of bacteria on the surface of the eye. These bacteria serve as potential sources for post-operative infection. One commonly used method is the administration of antibiotic drops 3 times: 1 hour prior to surgery at intervals of 5 minutes. Studies in the lab have shown that the preservative benzalkonium chloride 0.005%, part of the Zymar antibiotic drop preparation, allows the antibiotic to act more effectively than the antibiotic Vigamox, which does not include this preservative.

Comparison: The effect of Zymar antibiotic eye drops on conjunctival cultures compared to the effect of Vigamox on conjunctival cultures as measured by conjunctival cultures taken prior to treatment and then one hour after administration of eye drops 3 times, at 5 minute intervals.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 25 years of age or older
* Informed consent
* Likely to complete the entire course of the study

Exclusion Criteria:

* Contraindications or known sensitivity to any component of the study medications
* A subject on oral or topical antibiotics
* A subject that has a condition (i.e. an uncontrolled systemic disease) or is in a situation which, in the investigator's opinion, may put the subject at significant risk, may confound the trial results, or may interfere significantly with the subject's participation in the trial.
* Monocular subjects
* Contact lens wearers
* Subjects who regularly take eyedrops other than preservative free artificial tears
* A subject with an eye infection

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2006-06; Study Completion 2006-06

PRIMARY OUTCOMES:
Evidence of growth and number of colonies of bacteria on chocolate agar prior to antibiotic administration, t=0 hrs
Evidence of growth and number of colonies of bacteria on blood agar prior to antibiotic administration, t=0 hrs
Evidence of growth and number of colonies of bacteria on chocolate agar post-antibiotic administration, t=1 hr
Evidence of growth and number of colonies of bacteria on blood agar post-antibiotic administration, t=1 hr

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Raizman, B.A./M.D., Principal Investigator — Ophthalmic Consultants of Boston; Sandra Y Cho, B.A./M.D., Study Director — New England Eye Center/Tufts-New England Medical Center; Rahul Mandiga, B.S., Study Director — New England Eye Center/Tufts-New England Medical Center
Locations (1):
- Ophthalmic Consultants of Boston, Boston, Massachusetts, United States